CLINICAL TRIAL: NCT06367582
Title: Safety and Clinical Performance Assessment of Bone Cements and Injection Systems Used in Spine Surgery - A Post-Market Clinical Follow-Up
Brief Title: Spine Bone Cements Outcomes - Post Market Follow-up
Status: Recruiting | Type: Observational
Sponsor: Teknimed (Industry)
Responsible Party: Sponsor
Other Study IDs: CV01-TK-SPINE
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Vertebral Fracture; Compression Fracture; Osteoporotic Fractures
MeSH Terms: conditions — Spinal Fractures; Fractures, Compression; Osteoporotic Fractures | interventions — Vertebroplasty; Kyphoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (9):
- F20 VP: Vertebroplasty
  Interventions: Device: Vertebroplasty (VP)
- F20 KP: Kyphoplasty
  Interventions: Device: Kyphoplasty (KP)
- SPINEFIX VP: Vertebroplasty
  Interventions: Device: Vertebroplasty (VP)
- SPINEFIX KP: Kyphoplasty
  Interventions: Device: Kyphoplasty (KP)
- SPINEFIX PSA: Pedicular Screw Augmentation
  Interventions: Device: Pedicular Screw Augmentation (PSA)
- HIGH V+ VP: Vertebroplasty
  Interventions: Device: Vertebroplasty (VP)
- HIGH V+ KP: Kyphoplasty
  Interventions: Device: Kyphoplasty (KP)
- OPACITY+ VP: Vertebroplasty
  Interventions: Device: Vertebroplasty (VP)
- OPACITY+ KP: Kyphoplasty
  Interventions: Device: Kyphoplasty (KP)

INTERVENTIONS:
Device: Vertebroplasty (VP) — Vertebroplasty is a procedure in which a special medical-grade cement mixture is injected into a fractured vertebra to relieve pain
  Groups: F20 VP; HIGH V+ VP; OPACITY+ VP; SPINEFIX VP
Device: Kyphoplasty (KP) — Kyphoplasty is a procedure in which a special medical-grade cement mixture is injected into a fractured vertebra to relieve pain
  Groups: F20 KP; HIGH V+ KP; OPACITY+ KP; SPINEFIX KP
Device: Pedicular Screw Augmentation (PSA) — Pedicular Screw Augmentation is a procedure in which a special medical-grade cement mixture is injected into pedicular screws in order to augment fixation strength
  Groups: SPINEFIX PSA

SUMMARY:
A Post-Market Clinical Follow-Up (PMCF) Study to collect clinical data on safety and performance of all TEKNIMED Spine range of products: SPINEFIX, HIGH V+, OPACITY+ and F20 bone cements and mixing and injection systems, and all their private labels.

TEKNIMED bone cements are legacy products, some marketed for more than 10 years. Their performance and safety have already been demonstrated by Post-Market Surveillance and previous clinical studies. The current Post-Market Clinical Follow-Up study aims to confirm these claims by collecting data in a "real-life" setting.

The study is a retrospective and prospective global, single arm, non-controlled, multicentric, prospective observational study. Patients will be followed as per local standard medical care of the sites.

DETAILED DESCRIPTION:
It is admitted that:

* Cementoplasty procedures such as vertebroplasty and kyphoplasty are recommended in the treatment of painful vertebral compression fractures, due to their efficiency and safety
* These mini-invasive procedures, where bone cement is injected into a partially collapsed vertebral body, are used to reduce pain and to provide mechanical stability
* In most patients, a rapid pain relief and an increase in mobility and quality of life are obtained
* Serious complications from bone cements leaks and adjacent vertebral fractures can be observed but remain rather rare
* The use of spinal cement in pedicle screw augmentation procedures can be relevant to increase the strength of the screw fixation in the bone, particularly in osteoporotic patients.

TEKNIMED has developed several bone cements currently used in vertebroplasty and kyphoplasty procedures in the treatment of vertebral weakness. Among those, one cement is also used in pedicle screw augmentation procedures.

With the increasing use of these procedures, there is a need of real-life safety and efficacy data on the bone cements.

This retro-prospective study is performed to confirm the safety and performance of TEKNIMED spine bone cements in their current clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Be willing to sign an informed consent approved by Ethic Committee (when applicable) or not being opposed to the use of their clinical data in the study

  o For prospective inclusion:
* Be considered for treatment with one of the TEKNIMED Spine Range cement comprised in this study

  o For retrospective inclusion:
* Have undergone a surgery with a TEKNIMED Spine Range cement between the 1st of January 2016 and the date of the site initiation visit.
* Be informed of the study and not being opposed to the use of their clinical data in the study or be willing to sign an informed consent during the first follow-up visit following the site initiation (when applicable).

Exclusion Criteria:

Patients presenting one of the following conditions will not be included (contraindications per IFU):

* Procedures other than those stated in the INDICATIONS section
* Coagulation disorders, or severe cardiopulmonary disease
* Unstable vertebral fractures
* Compromise of the vertebral body or of the pedicle walls
* Hypersensitivity or allergy to one of the constituents of the product
* Patient clearly improving on more conservative treatment
* Prophylactic use in spinal metastatic or osteoporotic patients with no evidence of acute fracture
* Paediatric patients and pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from painful vertebral compression fractures resulting from osteoporosis, benign or malignant lesions, or of traumatic origin
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2029-09-04 (Estimated); Study Completion 2039-09-30 (Estimated)

PRIMARY OUTCOMES:
Alleviation of Pain | 24 months
  Pain evaluated by Visual Analogue Scale (VAS): on a scale of 0 to 10, with 0 being no pain and 10 being the most severe pain at the Baseline and at the Follow-up visits

SECONDARY OUTCOMES:
Restoration of quality of life | 24 months
  Evaluated through short questions : Oswestry Disability Index (ODI score)
Patient satisfaction | 24 months
  Evaluated through short questions :
  A. Are you satisfied with your surgery? Yes/No/Without opinion B. Has your health improved? Yes/Stable/No C. Given the results, would you accept this intervention again? Yes/No/Without opinion
Stabilization of vertebrae | 24 months
  Radiographic imaging
Adverse events | 10 years
  All adverse events occured during surgery and through study completion
Antalgic Consumption | 24 months
  Antalgic consumption and the drug type at the Baseline and at the Follow-up visits

CONTACTS AND LOCATIONS:
Locations (12):
- France (5):
  - CHU HautePierre, Strasbourg, Bas-Rhin
  - Pôle Rachis Hôpital Privé d'Eure et Loir, Mainvilliers, Eure et Loir
  - Hôpital Toulouse Purpan, Toulouse, Haute Garonne
  - Pôle Sud Santé, Le Mans, Sarthe
  - Centre Hospitalier Métropole Savoie, Chambéry, Savoie
- Hospitale Cruz Vermelha Portuguesa, Lisbon, Portugal
- Spain (5):
  - Clínica Teknon Instituto de neurociencias, Barcelona
  - Hospital Neurotraumatologico, Granada
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Fundacio Assistencial Mutua de Terrassa - Edifici Estació, Terrassa
  - Hospital de Zafra, Zafra
- Institute of Traumatology and Orthopaedics, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: No